CLINICAL TRIAL: NCT00379171
Title: The Importance of Complementary Feeding on Growth, Nutritional Status and Markers for Disease. An Intervention Study With Milk Types and LC-PUFA Supplements in 9- to 12-Month-Old Infants
Brief Title: Milk Types and Fish Oil in 9- to 12-Month-Old Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Anjo A/S (Unknown)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: KF 02-014/03; D-74
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Obesity; Metabolic Syndrome; Growth; Blood Pressure; Cardiovascular Disease
Keywords: Children; Complementary feeding; Breast feeding; Cow's milk; Formula; Protein; LCPUFA; Fish oil; Lipid profile; Intestinal inflammation; Intestinal microbiota
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Cardiovascular Diseases; Breast Feeding | interventions — Milk; Fish Oils; Food, Formulated

INTERVENTIONS:
Behavioral: Cow's milk with fish oil
Behavioral: Cow's milk without fish oil
Behavioral: Formula with fish oil
Behavioral: Formula without fish oil

SUMMARY:
The objective of this intervention study is to examine the effect of whole cow's milk versus infant formula as primary milk sources with or without supplements of n-3 LCPUFA for growth, nutritional status, development, risk factors for later diseases and the impact on the intestinal microbiota and inflammation in 9 - 12 months old infants.

ELIGIBILITY:
Inclusion Criteria:

* Singleton infants
* Born >= 37 wk of gestation
* Birth weight > 2500g
* >= 5th percentile for gestational age
* A 5-min Apgar score >= 7
* Daily consumption of cow's milk or formula

Exclusion Criteria:

* No major complications at birth or in fetal life
* No chronic diseases

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100
Dates: Start 2003-05; Study Completion 2004-03

PRIMARY OUTCOMES:
Growth
Body composition (weight, length, knee-heel-length, waist, head, and arm circumference, skin fold measurements).
IGF-I
IGFBP-3
Insulin - glucose metabolism (HOMA index).
Urea Nitrogen
Albumin
C-peptide
Amino Acids
Erythrocyte fatty acid composition
Blood pressure
Lipid Profile
Heart Rate Variability (HRV)
In vitro cytokine production from stimulated full blood (IL-10, IFN-gamma, TNF-alpha)
Plasma IgE, IL-2R, and CRP

SECONDARY OUTCOMES:
Plasma concentrations of cholesterol and triglycerides
Allergy status
Cognitive test ("The infant means-end problem solving test")
Iron status (hemoglobin, ferritin and transferrin receptors)
Feces samples: Calprotectin, IgA and composition of the intestinal microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Dr Med Sci, Study Chair — Institute of Human Nutrition, Rolighedsvej 30, DK-1958 Frederiksberg C, Denmark

REFERENCES:
- [Result] Lauritzen L, Christensen JH, Damsgaard CT, Michaelsen KF. The effect of fish oil supplementation on heart rate in healthy Danish infants. Pediatr Res. 2008 Dec;64(6):610-4. doi: 10.1203/PDR.0b013e318186e5c5. PMID 18679165
- [Result] Nielsen S, Nielsen DS, Lauritzen L, Jakobsen M, Michaelsen KF. Impact of diet on the intestinal microbiota in 10-month-old infants. J Pediatr Gastroenterol Nutr. 2007 May;44(5):613-8. doi: 10.1097/MPG.0b013e3180406a11. PMID 17460496
- [Result] Damsgaard CT, Lauritzen L, Kjaer TM, Holm PM, Fruekilde MB, Michaelsen KF, Frokiaer H. Fish oil supplementation modulates immune function in healthy infants. J Nutr. 2007 Apr;137(4):1031-6. doi: 10.1093/jn/137.4.1031. PMID 17374672
- [Result] Damsgaard CT, Schack-Nielsen L, Michaelsen KF, Fruekilde MB, Hels O, Lauritzen L. Fish oil affects blood pressure and the plasma lipid profile in healthy Danish infants. J Nutr. 2006 Jan;136(1):94-9. doi: 10.1093/jn/136.1.94. PMID 16365065
- See also: Damsgaard CT, Schack-Nielsen L, Michaelsen KF, Fruekilde MB, Hels O, Lauritzen L. Fish oil affects blood pressure and the plasma lipid profile in healthy danish infants. J Nutr 2006;136:94-9. — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Citation&list_uids=16365065